CLINICAL TRIAL: NCT07181057
Title: Synergistic Effects of Green Tea Extract and Ginger Supplementation on Endurance Performance and Thermal Perception in Normal and Cold Environments: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study
Brief Title: Neurocognitive Effects of Meal Timing in a One-Meal-a-Day Regimen
Acronym: OMAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Süleyman Ulupınar, Associate Professor of Exercise Physiology, Erzurum Technical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ETU-OMAD-2025-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Fasting State; Cognitive Abilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Crossover) (Experimental): Arm Title: Morning Meal (08:00) Arm Type: Experimental Intervention: Other: One-meal-a-day (OMAD) Arm Description: Participants consume a single standardized isocaloric meal at 08:00. Neurocognitive outcomes (ERP, resting-state EEG, Stroop performance) are assessed during morning (before meal) and afternoon (approximately 6 hours post-meal) sessions.
  Arm Title: Midday Meal (12:30) Arm Type: Experimental Intervention: Other: One-meal-a-day (OMAD) Arm Description: Participants consume a single standardized isocaloric meal at 12:30. Neurocognitive outcomes (ERP, resting-state EEG, Stroop performance) are assessed during morning (before meal) and afternoon (approximately 6 hours post-meal) sessions.
  Arm Title: Evening Meal (18:00) Arm Type: Experimental Intervention: Other: One-meal-a-day (OMAD) Arm Description: Participants consume a single standardized isocaloric meal at 18:00. Neurocognitive outcomes (ERP, resting-state EEG, Stroop performance) are assessed during morning (before mea
  Interventions: Other: one-meal-a-day (OMAD)

INTERVENTIONS:
Other: one-meal-a-day (OMAD) — Arm Title: Morning Meal (08:00)
  Intervention: Other: One-meal-a-day (OMAD)
  Description: Participants consume a single isocaloric meal at 08:00.
  Arm Title: Midday Meal (12:30)
  Intervention: Other: One-meal-a-day (OMAD)
  Description: Participants consume a single isocaloric meal at 12:30.
  Arm Title: Evening Meal (18:00)
  Intervention: Other: One-meal-a-day (OMAD)
  Description: Participants consume a single isocaloric meal at 18:00.

SUMMARY:
Objectives: The purpose of this study is to examine how meal timing in a one-meal-a-day (OMAD) regimen influences neurocognitive outcomes.

Methods: Twelve cognitively active participants (academics, students, software engineers) will complete three randomized OMAD conditions, consuming a standardized isocaloric meal at 08:00, 12:30, or 18:00. ERPs will be recorded during a computerized Stroop task to evaluate peak amplitudes and latencies under congruent and incongruent conditions. Resting-state EEG will be measured under eyes-open and eyes-closed conditions. Behavioral performance on the Stroop task, including reaction time and accuracy, will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Male, 20 to 45 years of age

Right-handed

Normal or corrected-to-normal vision

Cognitively active individuals (academic staff, graduate students, or software/algorithm engineers)

Regular sleep-wake schedule during the week preceding the experiment

Ability to abstain from caffeine, alcohol, or psychoactive substances for at least 24 hours prior to each test session

Body mass index between 18.5 and 30 kg/m²

Exclusion Criteria:

History of neurological, psychiatric, metabolic, or sleep disorders

Current use of medications that affect the central nervous system

Shift work or irregular sleep patterns (verified by sleep diary)

Prior experience with one-meal-a-day dietary routines

Body mass index below 18.5 or above 30 kg/m²

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To minimize hormone-related variability in electroencephalography and event-related potential measures in this pilot crossover study, enrollment is limited to males.
Enrollment: 12 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Positive Peak Amplitude of Event-Related Potentials During Stroop - Congruent Trials | Day 1 Morning session (09:30-11:00, pre-meal) and Day 1 Afternoon session (14:30-16:00, ~6 hours post-meal). Each participant completes three separate test days (morning, midday, evening feeding), ≥48 hours apart.
  Maximum voltage deflection (µV) within 250-450 ms after stimulus onset at CP1, CP2, Pz, P3, O1, and O2 electrodes, recorded during congruent Stroop trials using a 32-channel EEG system.
Latency of Positive Peak of Event-Related Potentials During Stroop - Congruent Trials | Day 1 Morning session (09:30-11:00, pre-meal) and Day 1 Afternoon session (14:30-16:00, ~6 hours post-meal). Each participant completes three separate test days (morning, midday, evening feeding), ≥48 hours apart.
  Time point (ms) of maximum positive deflection within 250-450 ms after stimulus onset at CP1, CP2, Pz, P3, O1, and O2 electrodes.

SECONDARY OUTCOMES:
Resting-State EEG Absolute Power (Eyes-Open and Eyes-Closed) | Day 1 Morning session (09:30-11:00, pre-meal) and Day 1 Afternoon session (14:30-16:00, ~6 hours post-meal). Each participant completes three separate test days (morning, midday, evening feeding), ≥48 hours apart.
  Broadband spectral power (µV²) recorded at CP1, CP2, Pz, P3, O1, and O2 electrodes during standardized eyes-open and eyes-closed resting-state EEG.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University Sport Sciences Faculty, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No